CLINICAL TRIAL: NCT01993199
Title: Prospective Study: Deep Biopsy Via Endoscopic Submucosal Dissection in Upper GI Subepithelial Tumors
Brief Title: Deep Biopsy Via Endoscopic Submucosal Dissection in Upper GI Subepithelial Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Lee Hang Lak, Professor, Hanyang University Seoul Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: deep biopsy111
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Benign Neoplasm; Pathology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- deep biopsy (Active Comparator)
  Interventions: Procedure: deep biopsy via ESD technique

INTERVENTIONS:
Procedure: deep biopsy via ESD technique

SUMMARY:
Upper gastrointestinal subepithelial tumors are frequently encountered during esophagogastroduodenoscopy. Treatment plans for subepithelial tumors are determined by algorithms based on endoscopic ultrasonography images. However, endoscopic ultrasonography alone may not be able to diagnose and evaluate upper gastrointestinal SETs with sufficient accuracy. Adequate tissue samples are required to increase the diagnostic accuracy of subepithelial tumors.

Deep biopsy is method that normal mucosa was dissected using enodsocpi submucosal dissection technique and multiple endoscopic biopsies were performed.

The investigators will perform deep biopsy in subepithelial tumor.

ELIGIBILITY:
Inclusion Criteria:

* patients with upper GI SETs

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the number of pathologic diagnosis of deep biopsy | within the 7 day

REFERENCES:
- [Derived] Tae HJ, Lee HL, Lee KN, Jun DW, Lee OY, Han DS, Yoon BC, Choi HS, Hahm JS. Deep biopsy via endoscopic submucosal dissection in upper gastrointestinal subepithelial tumors: a prospective study. Endoscopy. 2014 Oct;46(10):845-50. doi: 10.1055/s-0034-1377627. Epub 2014 Aug 11. PMID 25111136